CLINICAL TRIAL: NCT03623555
Title: Building Resilience Among Women: a Social Neuroscience Approach for the Prevention of Intimate Partner Violence Consequences
Brief Title: Applied Social Neuroscience: the Building Resilience Among Women Project
Acronym: BRAW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ximena Goldberg (Other)
Collaborators: La Caixa Foundation (Other); Universitat Autonoma de Barcelona (Other); Associació Catalana d'Universitats Públiques (Unknown)
Responsible Party: Sponsor-Investigator, Ximena Goldberg, Principal Investigator, Corporacion Parc Tauli
Organization: Corporacion Parc Tauli (Other)
Other Study IDs: BRAW2018
Record Dates: First submitted 2018-07-23; First posted 2018-08-09 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Violence, Domestic; Stress Related Disorder; Depressive Disorder
Keywords: Stress regulation; Depression; Intimate partner violence; Resilience; Psychophysiology; Endocrine response; Risk factor
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood, saliva, hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- E-IPV: Women who have been exposed to intimate partner violence. Half of this group will also have a history of childhood maltreatment.
  Women will be assessed for behavioral performance during the Trier Social Stress Test, and salivary cortisol will be collected.
  Interventions: Behavioral: Trier Social Stress Test; Biological: Salivary cortisol
- NE-IPV: Women who have never been exposed to intimate partner violence. Half of this group will also present a diagnosis of Major Depressive Disorder.
  Women will be assessed for behavioral performance during the Trier Social Stress Test, and salivary cortisol will be collected.
  Interventions: Behavioral: Trier Social Stress Test; Biological: Salivary cortisol

INTERVENTIONS:
Behavioral: Trier Social Stress Test — The participants are instructed to imagine having applied for their "dream job" and that they are now invited to a job interview. The TSST consists of three successive phases: (1) A preparation period (3min), (2) a free speech task in which the participants have to argue why they are the best candidate for the job they wish to apply for (5min), and (3) a mental arithmetic task in which participants have to sequentially subtract an odd two-digit number from an odd four-digit number (e.g., 17 from 2023; 5min). The two tasks are performed in front of a selection committee (two members), dressed in white lab coats, acting in a reserved manner and providing no facial or verbal feedback.
Biological: Salivary cortisol — Saliva samples will be obtained by means of Salivette collection devices before, 10 minutes after, and 30 minutes after the beginning of the TSST

SUMMARY:
Intimate partner violence (IPV) is the most common and alarming form of violence against women, affecting up to 25% of all women in Catalonia. It is a complex phenomenon that involves aspects of social interaction, cognitive-emotional processes, neurobiological alterations and cultural context. Using an integrative methodology, IPV will be approached as a form of chronic exposure to severe stress that alters the stress-response system of exposed women, affecting their capacity to cope with future everyday situations. Fortunately, coping strategies can be subject to change through learning mechanisms and thus the identification of vulnerabilities can help build resilience strategies that may have a long-lasting impression on women's healthy functioning.

It is proposed that the sustained exposure to violent social interactions impacts two key aspects of future behavior: i) altered psychosocial coping, and ii) enhanced emotional reactivity to acute stress. To test this hypothesis, the psychosocial and neurobiological response to common social acute stress will be analyzed among women with and without previous exposure to IPV. The Trier Social Stress Task (TSST) will be used, which is a valid test of acute stress that resembles the real life situation of a (mock) job interview. Based on a social neuroscience perspective, quantitative and qualitative measures will be used of cognitive performance, neuroendocrine activity and face-to-face interviews to obtain an integrative description of the response to the TSST that includes the personal narrative of the experience by women themselves.

Finally, the proposal will benefit from the fact that all participants will share the same experimental condition (the TSST), and this mock job interview will be used as the common reference point for a workshop about the difficulties and strengths put to test during a stressful situation. The focus of this workshop will be on raising awareness of such coping limitations and abilities that participants themselves will be able to identify. The results of this workshop will inform guidelines and recommendations for future work and prevention strategies, and participants will be invited to be an active part in our dissemination strategy

DETAILED DESCRIPTION:
The burden and prevalence of intimate partner violence (IPV) has helped recognized this issue as a global public health problem, one of particular interest in the field of mental health as women who suffer intimate partner violence present an increased prevalence of depression compared with non-exposed women. The devastating consequences of IPV on women's health have been attributed to an enduring impact of IPV on the stress system that has long-term consequences on the victim's quality of life and are mediated by changes in neuroendocrine system, particularly the hypothalamic-pituitary-adrenal (HPA) axis.

Despite the critical importance of this stress system, most research on IPV has merely evaluated basal HPA activity, leaving unanswered the question of responsiveness: do women previously exposed to IPV have difficulties when coping with new emotional situations? The activation of the stress system in response to novel stressful situations is a central matter as it reflects the person's capacity to respond to the changing demands that commonly occur at work and at home. Biases for threat have been linked to chronic stress and violence, and are associated with HPA axis activity.

Under these conditions, an altered stress response may have important consequences in women's future development. For example, a job interview could be a stressful circumstance that affected women may have to face after recovering from IPV. The performance during the interview (i.e. getting or losing the job opportunity) will largely depend on the person's vulnerability to emotionally stressful situations or, on the contrary, on the successful strategies women may present to cope with acute stress. The present proposal aims at identifying these learnt vulnerabilities and resilience resources among IPV-exposed women, using valid measures of psychosocial and neuroendocrine response to acute stress.

It is hypothesized that women exposed to IPV will present a profile of increased stress vulnerability characterized by: i) a sensitized HPA axis response to acute stress, and ii) a dysfunctional psychosocial response.

To test this hypothesis, a group of women with a history of IPV will be compared to a group of women without such history from the same community in order to: 1) Assess the long-term impact of IPV on the patterns of psychosocial coping (i.e. personal attitudes and perceptions, and selective attentional processing bias) and neuroendocrine response to acute stress, 2) Examine the association between IPV and an "increased vulnerability to stress profile" characterized by dysfunctional psychosocial and neuroendocrine responses to acute stress, 3) Identify the strategies used by resilient women (psychosocial schemes, neuroendocrine regulation) to cope with acute stress, and 4) Explore the value of the above findings to inform the development of prevention resources for IPV-exposed women and at-risk groups.

Procedures: Adult women will be recruited from the Primary attention unit and the Adults Mental Health Unit at the reference Hospital. Three main groups of women will be included: women exposed to intimate partner violence (E-IPV), women not exposed to IPV (NE-IPV), and not exposed to IPV with major depression disorder. This last group will provide a comparison group in relation to mental health disorders. Groups will be matched by age, socioeconomic position and educational level.

Sample size calculation: The task used to assess stress reactivity (Trier social stress task) reliably activates the HPA axis and triggers a two- to three-fold release of cortisol in about 70-80% of participants. Assuming an increase in hormones with the task of about 70% and a standard deviation of 30% of the mean, a sample size of 43 participants per group will be needed to detect differences among the two groups of half of this increase with a power of 0.80 and an alpha of 0.05. Therefore, the complete sample will include: i) the E-IPV group composed of 90 women, 43 of them with history of childhood abuse and 43 of them without such history, and ii) a NE-IPV group composed of 90 women, 43 of them healthy controls and 43 with a diagnosis of major depression disorder. Total sample size: 172 women.

Work plan: After identification of the participants according to the project's criteria, women will be contacted by a researcher and one interviewer will be assigned to each woman all through the assessment. The objectives and the activities of this study will be clearly differentiated from those of any assistance that participants may be receiving in other services. Women willing to receive a full laboratory and hair cortisol analysis will be referred for blood extraction and collection of hair sample. Assessments will be performed in two different days separated by a two-week period. On day one, participants will respond to the initial interview including demographics, clinical and physical information. On day two, participants will respond to a social stress task that will be followed by a post-task face-to-face interview. A saliva sample will be collected before the beginning of the task, again 10 minutes after the beginning of the task, and finally 30 minutes after the beginning of the task.

Data analysis: A detailed descriptive analysis will be run that includes the information from the initial interview and the neuroendocrine response trajectories during the TSST. With this information groups will be compared (E-IPV with and without childhood abuse, and NE-IPV with and without depression) to test for putative psychosocial and neurobiological differences at the level of stress response. These data will be analysed with standard statistical methods and the Statistical Package of Social Sciences (SPSS, Chicago) software.

Ethical considerations: Following WHO's recommendations, participants who come to the interview accompanied by their partners will not be included. No participant will be excluded on the basis of their ethnicity, religion or sexual orientation. Written informed consent (previously approved by the Ethics Committee) will be obtained after a full description of the study's aims and design. Participants will be informed of the confidentiality of their comments following data protection laws (European data protection law: 2016/679). Registry and use of information resulting from this study will follow the Declaration of Helsinki agreements and local laws on biomedical research (Law 14/2007 of Biomedical Research). The collected data will be identified by means of a code that guarantees the confidentiality of the information. The results obtained from the analysis of the sample will be dissociated from the personal data and the health information obtained. Biological samples will be stored under a collection located in the Hospital laboratories, from which the main researcher of the study will be the holder, and that will be registered in the National Registry of Biobanks.

ELIGIBILITY:
Inclusion Criteria for both groups:

* E-IPV group: - past history of at least 1 year of IPV exposure after the age of 18.

  * At least one year of established cessation of exposure to IPV
* Subgroup with childhood maltreatment: - history of childhood maltreatment before the age of 16.
* NE-IPV group: - no history of IPV lifetime

  * no history of childhood maltreatment
* Subgroup with major depression disorder: - Presence of major depression disorder in the last year

Two groups of women will be included: women exposed to IPV (E-IPV), and women not ex-posed to IPV (NE-IPV). Inclusion criteria for the E-IPV group: (Index of Spouse Abuse18,19; Woman Abuse Screening Tool20,21). Inclusion criteria for the NE-IPV group: no history of IPV or any other form of chronic exposure to violent behaviour. Exclusion criteria for both groups: inability to read or comprehend instructions, pregnancy, current use of steroid-based medications and/or presence of any endocrine alteration. Groups will be matched by age, socioeconomic position and educational level.

Exclusion Criteria (both groups):

* Age under 25 or over 45 years old.
* Endocrine alteration, including steroid-based illness/medication
* Pregnancy (last 6 months), current breast-feeding.
* Current disability or illness that may cause inability to read or comprehend instructions

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population under study are women between 25 and 45 years of age
Sampling Method: Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Salivary cortisol | Recovery after acute stress response experiment (TSST): 45 minutes
  Salivary cortisol concentration levels

SECONDARY OUTCOMES:
Behavioral response | Recovery after acute stress response experiment (TSST): 45 minutes
  Behavioral performance during acute stress response experiment (TSST)

CONTACTS AND LOCATIONS:
Locations (1):
- Parc Taulí University Hospital, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li SH, Graham BM. Why are women so vulnerable to anxiety, trauma-related and stress-related disorders? The potential role of sex hormones. Lancet Psychiatry. 2017 Jan;4(1):73-82. doi: 10.1016/S2215-0366(16)30358-3. Epub 2016 Nov 15. PMID 27856395
- [Background] Kuehner C. Why is depression more common among women than among men? Lancet Psychiatry. 2017 Feb;4(2):146-158. doi: 10.1016/S2215-0366(16)30263-2. Epub 2016 Nov 15. PMID 27856392
- [Background] Inslicht SS, Marmar CR, Neylan TC, Metzler TJ, Hart SL, Otte C, McCaslin SE, Larkin GL, Hyman KB, Baum A. Increased cortisol in women with intimate partner violence-related posttraumatic stress disorder. Psychoneuroendocrinology. 2006 Aug;31(7):825-38. doi: 10.1016/j.psyneuen.2006.03.007. Epub 2006 May 23. PMID 16716530
- [Background] Pinna KL, Johnson DM, Delahanty DL. PTSD, comorbid depression, and the cortisol waking response in victims of intimate partner violence: preliminary evidence. Anxiety Stress Coping. 2014 May;27(3):253-69. doi: 10.1080/10615806.2013.852185. Epub 2013 Nov 28. PMID 24283327
- [Background] Belda X, Fuentes S, Daviu N, Nadal R, Armario A. Stress-induced sensitization: the hypothalamic-pituitary-adrenal axis and beyond. Stress. 2015;18(3):269-79. doi: 10.3109/10253890.2015.1067678. Epub 2015 Aug 17. PMID 26300109
- [Background] Oram S, Khalifeh H, Howard LM. Violence against women and mental health. Lancet Psychiatry. 2017 Feb;4(2):159-170. doi: 10.1016/S2215-0366(16)30261-9. Epub 2016 Nov 15. PMID 27856393
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Frisch JU, Hausser JA, Mojzisch A. The Trier Social Stress Test as a paradigm to study how people respond to threat in social interactions. Front Psychol. 2015 Feb 2;6:14. doi: 10.3389/fpsyg.2015.00014. eCollection 2015. PMID 25698987
- [Derived] Goldberg X, Espelt C, Palao D, Nadal R, Armario A. Adaptability to acute stress among women survivors of intimate partner violence: protocol for a mixed-methods cross-sectional study in a laboratory setting (BRAW study). BMJ Open. 2020 Oct 1;10(10):e036561. doi: 10.1136/bmjopen-2019-036561. PMID 33004387
- See also: World Health Organization. Global and regional estimates of violence against women: prevalence and health effects of intimate partner violence and non-partner sexual violence — http://apps.who.int/iris/bitstream/handle/10665/85239/9789241564625_eng.pdf;jsessionid=0D5290C5C1A82D611EC6B26848B7FA66?sequence=1
- See also: Catalan Institute of Women. Violence against women, data from Catalonia — http://dones.gencat.cat/web/.content/03_ambits/docs/vm_l900_2015_resumdades.pdf